CLINICAL TRIAL: NCT03905655
Title: Randomized Double-Blind Study of Nitazoxanide Compared to Placebo in Subjects With HBeAG-Negative Chronic Hepatitis B Virologically Suppressed for at Least Twelve Months on Tenofovir Disoproxil Fumarate, Tenofovir Alafenamide or Entecavir
Brief Title: Study of Nitazoxanide Compared to Placebo in Subjects With HBeAG-Negative Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM08-2001
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Patients are randomized 1:1:1:1 (12 subjects per group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Placebo Comparator): Three placebo tablets administered orally twice daily with food in addition to continuing TDF, TAF or ETV therapy
  Interventions: Drug: Placebo Oral Tablet
- Group 2 (Active Comparator): Two 300 mg NTZ tablets and one placebo tablet administered orally in the morning and three placebo tablets in the evening in addition to continuing TDF, TAF or ETV therapy
  Interventions: Drug: Placebo Oral Tablet; Drug: Nitazoxanide
- Group 3 (Active Comparator): Two 300 mg NTZ tablets and one placebo tablet administered orally twice daily with food in addition to continuing TDF, TAF or ETV therapy
  Interventions: Drug: Placebo Oral Tablet; Drug: Nitazoxanide
- Group 4 (Active Comparator): Three 300 mg NTZ tablets administered orally twice daily with food in addition to continuing TDF, TAF or ETV therapy
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Placebo Oral Tablet — Number of placebo tablets administered orally depends on the arm
  Arms: Group 1; Group 2; Group 3
Drug: Nitazoxanide — Number of Nitazoxanide 300 mg extended release tablets administered orally depends on the arm
  Other Names: NTZ, NT-300
  Arms: Group 2; Group 3; Group 4

SUMMARY:
This randomized controlled trial is designed to evaluate safety, effectiveness and pharmacokinetic-pharmacodynamic (PK/PD) relationships associated with three different Nitazoxanide (NTZ) treatment regimens added to Tenofovir Disoproxil Fumarate (TDF), Tenofovir Alafenamide (TAF) or Entecavir (ETV) in treating Chronic Hepatitis B (CHB).

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 21 years
2. CHB virus infection (serum HBsAg-positive for at least 6 months or serum HBsAg-positive and negative immunoglobulin M (IgM) antibodies to Hepatitis B Virus (HBV) core antigen (IgM anti-HBc))
3. Hepatitis B e Antigen (HBeAg) negative
4. Virologically suppressed (HBV DNA less than the lower limit of quantitation) for at least 12 months on Tenofovir Disoproxil Fumarate (TDF), Tenofovir Alafenamide (TAF) or Entecavir (ETV) therapy
5. Quantitative HBsAg greater than 100 IU/mL
6. Alanine Aminotransferase (ALT) below 1.5 times the upper limit of normal
7. Able to comply with the study requirements

Exclusion Criteria:

1. Unable to take oral medications
2. Females who are pregnant, breast-feeding or not using birth control. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an intrauterine device (IUD), or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. In addition, female subjects should have a baseline pregnancy test and should agree to continue an acceptable method of birth control for the duration of the study (including follow-up) if sexually active.
3. Any investigational drug therapy within 30 days prior to enrollment
4. Other causes of liver disease
5. Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis D virus (HDV) based on an enzyme immunoassay (EIA)
6. History of alcoholism or with an alcohol consumption of greater than 40 g per day
7. Clinically unstable
8. Any concomitant condition that, in the opinion of the investigator would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed
9. History of hypersensitivity or intolerance to NTZ or any of the excipients comprising the NTZ tablets
10. Hepatocellular carcinoma
11. Decompensated liver disease including history of ascites, bleeding esophageal varices, portal hypertension or hepatic encephalopathy
12. FibroScan® score greater than 11 or history of cirrhosis on liver biopsy
13. Creatinine clearance <65 ml/minute (by the Cockcroft-Gault equation using ideal body weight)
14. History of clinically relevant psychiatric disease, seizures, central nervous system dysfunction, severe pre-existing cardiac, renal, pathologic bone fracture or other risk factors for osteoporosis, hematological disease or medical illness that in the investigator's opinion might interfere with therapy
15. Malignant disease within 3 years of trial entry
16. Rheumatological conditions, inflammatory bowel disease or psoriasis requiring or anticipated to require biological/immunosuppressive therapies
17. Subjects taking or anticipated to need medications considered to be major CYP2C8 substrates

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 13 | 13 | 11 | 14
Completed | 12 | 13 | 10 | 13
Not Completed | 1 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All subjects receiving at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 13 | 13 | 11 | 14 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (9.23) | 52.7 (9.17) | 47.7 (7.24) | 52.0 (10.35) | 49.8 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 3
  Male | 12 | 12 | 10 | 14 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 13 | 9 | 14 | 49
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 13 | 13 | 11 | 14 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 13 | 13 | 11 | 14 | 51
Quantitative HBsAg [Mean (Standard Deviation); unit: log10 IU/mL] | 3.1 (0.50) | 3.0 (0.45) | 3.0 (0.34) | 2.8 (0.51) | 3.0 (0.47)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Quantitative Hepatitis B Surface Antigen (qHBsAg)
Description: Mean change in quantitative Hepatitis B Surface Antigen (qHBsAg) from Baseline
Time Frame: Baseline to 12 weeks
Population: All subjects who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 12 | 13 | 10 | 13
log10 IU/mL | 0.0 (0.13) | 0.0 (0.90) | 0.0 (0.06) | 0.0 (0.10)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 2: Comparison: Group 1 vs Group 3; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 3: Comparison: Group 1 vs Group 4; Test type: Superiority; p = 1.000, t-test, 2 sided

2. Secondary Outcome: Sustained HBsAg Loss With Suppression of HBV DNA for 24 Weeks After the End of Treatment
Description: Proportion of participants with sustained HBsAg loss with suppression of HBV DNA for 24 weeks after the end of treatment
Time Frame: Baseline to 24 weeks after the end of treatment
Population: All participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 13 | 13 | 11 | 14
Participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 vs Group 3; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 vs Group 4; Test type: Superiority; p = 1.000, Fisher Exact

3. Secondary Outcome: Change in Quantitative Hepatitis B Surface Antigen (qHBsAg) From Baseline to Different Time Points on Treatment
Description: Change in mean Quantitative Hepatitis B Surface Antigen (qHBsAg) from Baseline to Day 3, Week 1, Week 2, Week 4, and Week 8
Time Frame: 8 weeks
Population: All participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 13 | 13 | 11 | 14
log10 IU/mL
  Day 3 | 0.0 (0.04) | 0.0 (0.08) | 0.0 (0.04) | 0.0 (0.06)
  Week 1 | 0.0 (0.06) | 0.0 (0.05) | 0.0 (0.04) | 0.0 (0.05)
  Week 2 | 0.0 (0.05) | 0.0 (0.11) | 0.0 (0.04) | 0.1 (0.05)
  Week 4 | 0.0 (0.08) | 0.0 (0.09) | 0.0 (0.05) | 0.1 (0.07)
  Week 8 | 0.0 (0.06) | 0.0 (0.14) | -0.1 (0.07) | 0.0 (0.10)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Comparison of Day 3 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Comparison of Week 1 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Comparison of Week 2 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Comparison of Week 4 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Comparison of Week 8 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 6: Comparison: Group 1 vs Group 3; Comparison of Day 3 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 7: Comparison: Group 1 vs Group 3; Comparison of Week 1 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 8: Comparison: Group 1 vs Group 3; Comparison of Week 2 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 9: Comparison: Group 1 vs Group 3; Comparison of Week 4 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 10: Comparison: Group 1 vs Group 3; Comparison of Week 8 values; Test type: Superiority; p = 0.001, t-test, 2 sided
Statistical Analysis 11: Comparison: Group 1 vs Group 4; Comparison of Day 3 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 12: Comparison: Group 1 vs Group 4; Comparison of Week 1 values; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 13: Comparison: Group 1 vs Group 4; Comparison of Week 2 values; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 14: Comparison: Group 1 vs Group 4; Comparison of Week 4 values; Test type: Superiority; p = 0.002, t-test, 2 sided
Statistical Analysis 15: Comparison: Group 1 vs Group 4; Comparison of Week 8 values; Test type: Superiority; p = 1.000, t-test, 2 sided

4. Secondary Outcome: Hepatitis B Surface Antigen (HBsAg) Loss
Description: Proportion of participants with HBsAg loss defined as quantitative HBsAg below the lower limit of quantitation at Day 3, Week 1, Week 2, Week 4, Week 8, and Week 12
Time Frame: 12 weeks
Population: All participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 13 | 13 | 11 | 14
Participants
  Day 3 | 0 | 0 | 0 | 0
  Week 1 | 0 | 0 | 0 | 0
  Week 2 | 0 | 0 | 0 | 0
  Week 4 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0
  Week 12 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 7: Comparison: Group 1 vs Group 3; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 8: Comparison: Group 1 vs Group 3; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 9: Comparison: Group 1 vs Group 3; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 10: Comparison: Group 1 vs Group 3; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 11: Comparison: Group 1 vs Group 3; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 12: Comparison: Group 1 vs Group 3; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 13: Comparison: Group 1 vs Group 4; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 14: Comparison: Group 1 vs Group 4; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 15: Comparison: Group 1 vs Group 4; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 16: Comparison: Group 1 vs Group 4; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 17: Comparison: Group 1 vs Group 4; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 18: Comparison: Group 1 vs Group 4; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact

5. Secondary Outcome: Hepatitis B Surface Antigen (HBsAg) Seroconversion
Description: Proportion of participants with hepatitis B surface antigen (HBsAg) seroconversion defined as HBsAg loss and gain of anti-hepatitis B antibodies at Day 3, Week 1, Week 2, Week 4, Week 8, and Week 12
Time Frame: 12 weeks
Population: All participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 13 | 13 | 11 | 14
Participants
  Day 3 | 0 | 0 | 0 | 0
  Week 1 | 0 | 0 | 0 | 0
  Week 2 | 0 | 0 | 0 | 0
  Week 4 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0
  Week 12 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 7: Comparison: Group 1 vs Group 3; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 8: Comparison: Group 1 vs Group 3; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 9: Comparison: Group 1 vs Group 3; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 10: Comparison: Group 1 vs Group 3; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 11: Comparison: Group 1 vs Group 3; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 12: Comparison: Group 1 vs Group 3; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 13: Comparison: Group 1 vs Group 4; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 14: Comparison: Group 1 vs Group 4; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 15: Comparison: Group 1 vs Group 4; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 16: Comparison: Group 1 vs Group 4; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 17: Comparison: Group 1 vs Group 4; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 18: Comparison: Group 1 vs Group 4; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact

6. Secondary Outcome: Hepatitis B Virus DNA Suppression
Description: Proportion of participants with hepatitis B virus DNA suppression defined as hepatitis B virus DNA below the lower limit of quantitation (20 IU/mL) at Day 3, Week 1, Week 2, Week 4, Week 8, and Week 12
Time Frame: 12 weeks
Population: All participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 13 | 13 | 11 | 14
Participants
  Day 3 | 13 | 13 | 11 | 13
  Week 1 | 13 | 12 | 11 | 14
  Week 2 | 13 | 12 | 11 | 13
  Week 4 | 13 | 12 | 11 | 13
  Week 8 | 13 | 12 | 11 | 14
  Week 12 | 13 | 13 | 11 | 13
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 7: Comparison: Group 1 vs Group 3; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 8: Comparison: Group 1 vs Group 3; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 9: Comparison: Group 1 vs Group 3; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 10: Comparison: Group 1 vs Group 3; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 11: Comparison: Group 1 vs Group 3; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 12: Comparison: Group 1 vs Group 3; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 13: Comparison: Group 1 vs Group 4; Comparison of Day 3 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 14: Comparison: Group 1 vs Group 4; Comparison of Week 1 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 15: Comparison: Group 1 vs Group 4; Comparison of Week 2 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 16: Comparison: Group 1 vs Group 4; Comparison of Week 4 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 17: Comparison: Group 1 vs Group 4; Comparison of Week 8 values; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 18: Comparison: Group 1 vs Group 4; Comparison of Week 12 values; Test type: Superiority; p = 1.000, Fisher Exact

7. Secondary Outcome: Change in Fibrosis-4 (FIB-4) Score
Description: Mean change in Fibrosis-4 (FIB-4) score from Baseline to Week 1, Week 2, Week 4, Week 8, and Week 12. FIB-4 score is calculated as (age in years * Aspartate aminotransferase (AST) in U/L)/(platelet count in 10^9 U/L * square root of alanine aminotransferase (ALT) in U/L). FIB-4 scores under 1.45 have a negative predictive value of 90% for advanced fibrosis (better outcome) and FIB-4 scores >3.25 have a positive predictive value of 65% for advanced fibrosis (worse outcome). See Sterling RK, Lissen E, Clumeck N, et. al. Development of a simple noninvasive index to predict significant fibrosis patients with HIV/HCV co-infection. Hepatology 2006;43:1317-1325.
Time Frame: 12 weeks
Population: All participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: FIB-4 Score
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 12 | 13 | 10 | 13
FIB-4 Score
  Week 1 | -1.7 (0.88) | -2.8 (0.97) | -2.9 (2.68) | -2.0 (0.86)
  Week 2 | -1.4 (1.08) | -2.8 (1.06) | -2.9 (2.61) | -1.8 (0.88)
  Week 4 | -1.7 (0.88) | -2.9 (1.03) | -2.9 (2.81) | -1.8 (1.07)
  Week 8 | -1.7 (1.00) | -2.9 (1.05) | -2.8 (2.67) | -2.1 (0.91)
  Week 12 | 0.0 (0.57) | -1.2 (1.06) | -1.0 (1.51) | -0.8 (0.76)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Comparison of Week 1 values; Test type: Superiority; p = 0.006, t-test, 2 sided
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Comparison of Week 2 values; Test type: Superiority; p = 0.003, t-test, 2 sided
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Comparison of Week 4 values; Test type: Superiority; p = 0.004, t-test, 2 sided
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Comparison of Week 8 values; Test type: Superiority; p = 0.006, t-test, 2 sided
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Comparison of Week 12 values; Test type: Superiority; p = 0.002, t-test, 2 sided
Statistical Analysis 6: Comparison: Group 1 vs Group 3; Comparison of Week 1 values; Test type: Superiority; p = 0.141, t-test, 2 sided
Statistical Analysis 7: Comparison: Group 1 vs Group 3; Comparison of Week 2 values; Test type: Superiority; p = 0.081, t-test, 2 sided
Statistical Analysis 8: Comparison: Group 1 vs Group 3; Comparison of Week 4 values; Test type: Superiority; p = 0.160, t-test, 2 sided
Statistical Analysis 9: Comparison: Group 1 vs Group 3; Comparison of Week 8 values; Test type: Superiority; p = 0.184, t-test, 2 sided
Statistical Analysis 10: Comparison: Group 1 vs Group 3; Comparison of Week 12 values; Test type: Superiority; p = 0.046, t-test, 2 sided
Statistical Analysis 11: Comparison: Group 1 vs Group 4; Comparison of Week 1 values; Test type: Superiority; p = 0.379, t-test, 2 sided
Statistical Analysis 12: Comparison: Group 1 vs Group 4; Comparison of Week 2 values; Test type: Superiority; p = 0.308, t-test, 2 sided
Statistical Analysis 13: Comparison: Group 1 vs Group 4; Comparison of Week 4 values; Test type: Superiority; p = 0.794, t-test, 2 sided
Statistical Analysis 14: Comparison: Group 1 vs Group 4; Comparison of Week 8 values; Test type: Superiority; p = 0.297, t-test, 2 sided
Statistical Analysis 15: Comparison: Group 1 vs Group 4; Comparison of Week 12 values; Test type: Superiority; p = 0.007, t-test, 2 sided

8. Secondary Outcome: Change in FibroScan Score
Description: Mean change in FibroScan score from Baseline to end of treatment. Fibroscan is a kind of liver elastography measuring liver stiffness in kilopascals (kPa). Higher results are consistent with liver disease (worse outcome).
Time Frame: Baseline to end of treatment
Population: All participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: kilopascals (kPa)
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 5 | 3 | 4 | 3
kilopascals (kPa) | 0.0 (1.41) | 2.0 (1.73) | 0.0 (0.82) | 1.3 (1.53)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.123, t-test, 2 sided
Statistical Analysis 2: Comparison: Group 1 vs Group 3; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 3: Comparison: Group 1 vs Group 4; Test type: Superiority; p = 0.266, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/11 | 1/14
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/13 | 0/11 | 1/14
Other Adverse Events (participants affected / at risk) | 10/13 | 10/13 | 11/11 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=13) | Group 2 (N=13) | Group 3 (N=11) | Group 4 (N=14)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mixed hepatocellular cholangiocarcinoma (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=13) | Group 2 (N=13) | Group 3 (N=11) | Group 4 (N=14)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scleral discolouration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (4) | 2 (2) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hunger (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (2) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 2 (2) | 8 (8) | 8 (10) | 11 (11)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was a pilot study with a small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT03905655/Prot_SAP_000.pdf